CLINICAL TRIAL: NCT03547817
Title: Intermittent Negative Pressure to Improve Blood Flow in Patients With Peripheral Artery Disease. An Experimental Study to Investigate the Optimal Pulse Pressure Regime to Improve Blood Flow.
Brief Title: Intermittent Negative Pressure to Improve Blood Flow in Patients With Peripheral Artery Disease: Optimal Pulse Pressure Regime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Otivio AS (Industry)
Responsible Party: Principal Investigator, Jonny Hisdal, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SD0321063
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication; Lower Extremity Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimal negative pulse pressure regime (Experimental): The equipment for physiological measurements will be attached to the patient, and the foot will then be placed in the pressure chamber of the intermittent negative pressure device. The device induces pulses of 10 sec negative pressure, and 7 sec of atmospheric pressure. Pressure levels of 0 mmHg, -10 mmHg, -20 mmHg, -40 mmHg and -60 mmHg will be tested, with washout periods of 5 minutes between the different pressure levels. The order of the different negative pressure levels will be randomized to avoid causal interference.
  Interventions: Device: Intermittent negative pressure device

INTERVENTIONS:
Device: Intermittent negative pressure device — Pressure levels of 0 mmHg, -10 mmHg, -20 mmHg, -40 mmHg and -60 mmHg will be tested, with washout periods of 5 minutes between the different pressure levels

SUMMARY:
Recent studies have shown that applying intermittent negative pressure (INP) with short negative pressure (-40 mmHg) pulses to the lower extremities increase arterial blood flow velocity and skin blood flow. However, the optimal magnitude of negative pressure to improve blood flow is not known, and needs further investigation. Peripheral arterial blood flow velocity, skin blood flow and skin temperature in the foot will be recorded at different levels of oscillating negative pressure to identify a pressure range which is practically, while at the same time induce clinically relevant changes in blood flow parameters. Heart rate and blood pressure will be recorded to monitor the effects on the central circulation.

DETAILED DESCRIPTION:
Cross sectional study design. The equipment for physiological measurements will be attached to the patient, and the foot will then be placed in the pressure chamber. The device induces pulses of 10 sec negative pressure, and 7 sec of atmospheric pressure. Pressure levels of 0 mmHg, -10mmHg, -20 mmHg, -40 mmHg and -60 mmHg will be tested.

Patients will be recruited from the out-patient clinic at Department of Vascular Surgery, Oslo University Hospital, Aker.

Inclusion criteria:

Diagnosed peripheral artery disease (PAD), Ankle-Brachial Index <0.9 Outcome measures:

Arterial blood flow: Ultrasound Doppler from peripheral arteries in the foot.

Skin blood flow: Laser Doppler to measure acral skin blood perfusion.

Skin temperature

Systemic blood pressure: Finger arterial pressure will continuously be acquired by a photoplethysmographic pressure recording device (Finometer).

Ankle brachial index

Pressure recordings inside the pressure chamber: Continuously monitoring of pressure within the pressure chamber using a digital differential manometer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed peripheral artery disease
* Ankle-Brachial Index <0.9

Exclusion Criteria:

* Incapable to make an informed consent
* Diagnosis of severe psychiatric disease
* Severe heart disease such as unstable angina pectoris, severe heart failure (NYHA IV), severe valve failure
* Systemic infection
* Use of vasoactive substances

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Arterial blood flow | At time of intervention
  Continuously Ultrasound Doppler measurements of the dorsalis pedis artery or tibialis posterior artery to monitor changes in arterial blood flow during 5 min sequences of intermittent negative pressure treatment. Pressure levels of 0, -10 mmHg, -20 mmHg, -40 mmHg and -60 mmHg will be tested. Systolic pressures in the arm and the ankle will be assessed before the intervention to describe the patients severity of disease.

SECONDARY OUTCOMES:
Skin blood flow | At time of intervention
  Continuously Laser Doppler measurements from the pulp of the first toe to monitor changes in acral skin perfusion during 5 min sequences of intermittent negative pressure treatment. Pressure levels of 0, -10 mmHg, -20 mmHg, -40 mmHg and -60 mmHg will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Jonny Hisdal, PhD, Principal Investigator — Department of Vascular diseases, Oslo University Hospital, Aker
Locations (1):
- Department of Vascular diseases, Oslo University Hosptital, Aker, Oslo, Norway